CLINICAL TRIAL: NCT05084183
Title: An Adaptive, Randomized, Controlled Trial Evaluating the Effectiveness of PermeaDerm® (PD) as Compared to Mepilex Ag® Used as Standard of Care in the Treatment of Adult and Pediatric Partial Thickness Burns.
Brief Title: Evaluation of the Effectiveness of PermeaDerm® (PD) as Compared to Mepilex Ag®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stedical Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST-2021-B001
Record Dates: First submitted 2021-09-16; First posted 2021-10-19 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Thermal Burn

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blinded, adaptive, controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: It is intended that blinded assessment of wounds will be performed at 14 days after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PermeaDerm® (Experimental): N=34 Participants will receive application of PermeaDerm® as outlined in Directions for Use
  Interventions: Device: PermeaDerm®
- Mepilex Ag® (Active Comparator): Participants will receive application of Mepilex Ag® as outlined in Directions for Use.
  Interventions: Device: Mepilex Ag

INTERVENTIONS:
Device: PermeaDerm® — Wound Management Device
  Arms: PermeaDerm®
Device: Mepilex Ag — Wound Dressing
  Arms: Mepilex Ag®

SUMMARY:
A total of 68 adult and pediatric patients who suffer from at least one discrete partial thickness thermal burn wound (Grade II) will be recruited. Subjects will be randomized (1:1) to either PermeaDerm® or Mepilex Ag®. Evaluations will occur at 7, 14 and 21 days with long term follow-up at 6 and 12 months.

DETAILED DESCRIPTION:
A total of 68 adult and pediatric patients who suffer from at least one discrete partial thickness thermal burn wound (Grade II) will be recruited from the clinical practices of the site Principal Investigators.

Participants and/or the Legally Authorized Representative (LAR) as appropriate will be fully informed regarding the conduct of the clinical trial including all potential risks and benefits.

All Participants must be consented, randomized (1:1) and treated within 72 hours of injury.

It is permissible for a Study Participant to be enrolled if they have more than one burn wound.

If more than one partial thickness burn is treated, the Investigator must indicate prior to randomization which wound is to be considered for primary analysis. This wound will be called the Primary Wound and is to be evaluated by a Blinded Assessor.

Additional partial thickness wounds must be treated with the same product to which the Study Participant was randomized and will be included in secondary analysis. These wounds are to be described as Secondary Wounds and are to be evaluated by the Unblinded Assessor.

Evaluations will occur at 7, 14 and 21 days with long term follow-up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included if all the following criteria are met.

1. Able to give informed consent and undergo treatment < 72 hours of injury (consent may be given by LAR as necessary);
2. Any adult or pediatric patient < 75 years of age;
3. Target burn to be at least one discrete partial thickness (second degree) thermal burns <20% total body surface area (TBSA) on anybody surface except the face;
4. Characteristics of treated wound (s) must be superficial to deep partial thickness wounds such that application of both PermeaDerm and Mepilex Ag is medically appropriate;
5. Agrees to abstain from the use of any other wound covering device for the duration of the study unless determined by the individual site Principal Investigator to be medically necessary;
6. Demonstrates the ability and willingness to follow the requirements of the protocol.

Exclusion Criteria:

Participants will be excluded if s/he meet any of the following criteria.

1. Pregnant or breastfeeding;
2. Target burn ≥ 20% TBSA;
3. Electrical burns, chemical burns, frostbite;
4. Treatment with silver sulfadiazine prior to presentation;
5. Has comorbidities and/or medications and/or health status that (at the discretion of the individual site Principal Investigator) could result in poor wound healing (some examples may include admission to intensive care unit, inhalation, or other significant burn associated conditions, uncontrolled and/or significant diabetes, peripheral vascular disease, active malignancy, autoimmune disease, smoking, drug abuse, renal failure, steroid usage.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Reepithelialization | 14 days
  Time to 100 percent- primary wound
Alternate therapy | 14 days
  Time to conversion to alternate therapy- primary wound

SECONDARY OUTCOMES:
Re-epithelialization | 14 days
  Percent reepithelialization primary and secondary Wounds
Alternate therapy | up to 12 Months
  Time to conversion to alternate therapy- secondary wounds
Adverse Events | 21 days
  Occurrence, duration, severity, seriousness, expectedness, and relationship of adverse events
Severity of pain | Up to 12 Months
  Wong-Backer Faces pain rating scale and in adults as measured by the Numerical Rating Scale (0-10);
Scar characteristics | 6 and 12 months
  Patient and Observer Scar Assessment Scale (POSAS)
Satisfaction with treatment | 6 and 12 months
  Brisbane Burn Scar Impact Profile (BBSIP)
Dressing Changes Required | Up to 21 Days
  Number

CONTACTS AND LOCATIONS:
Overall Officials: David Greenhalgh, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No